CLINICAL TRIAL: NCT00351143
Title: A Randomized, Open Label Comparative Study to Determine the Proportion of Asthma Patients on SERETIDE Diskus 50/250 mcg b.i.d. Achieving Total Control When Given Medication and Compliance Enhancement Training Compared to Those Receiving Medication Only
Brief Title: A Comparative Study To Determine If Motivating Asthma Education (Compliance Enhancement) Has An Effect On Asthma Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE104325
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: QoL; Asthma; asthma compliance enhancement; Salmeterol/fluticasone; Total control; SERETIDE; FEV1
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Interventional group: Period 2 (Experimental): Randomized subjects will receive salmeterol/fluticasone propionate 50/250 µg + 3 training sessions of compliance enhancement training in Period 2
  Interventions: Drug: salmeterol/fluticasone propionate 50/250 µg + 3 training sessions of compliance enhancement training
- Control group: Period 2 (Active Comparator): Randomized subjects will receive salmeterol/fluticasone propionate 50/250 µg in treatment Period 2
  Interventions: Drug: salmeterol/fluticasone propionate 50/250 µg
- Subjects receiving salmeterol/fluticasone propionate: Period 1 (Experimental): All subjects treated with salmeterol/fluticasone propionate 50/250 µg b.i.d without any other intervention will be included in Period 1
  Interventions: Drug: salmeterol/fluticasone propionate 50/250 µg

INTERVENTIONS:
Drug: salmeterol/fluticasone propionate 50/250 µg + 3 training sessions of compliance enhancement training — Salmeterol/fluticasone propionate 50/250 µg + 3 training sessions of compliance enhancement training will be provided to intervention group in Period 2.
  Arms: Interventional group: Period 2
Drug: salmeterol/fluticasone propionate 50/250 µg — Salmeterol/fluticasone propionate 50/250 µg will be administered to control group in Period 2
  Arms: Control group: Period 2; Subjects receiving salmeterol/fluticasone propionate: Period 1

SUMMARY:
This study will investigate whether study subjects with previously uncontrolled asthma treated with SERETIDE Diskus 50/250 CCI18781+GR33343 mcg twice a day can attain a level of Total Control of their condition and whether adherence to treatment can be enhanced by teaching the subjects. Two groups of equal size with identical medical treatment will be compared with each other, the test group receiving three training modules during study visits and the control group regular study visits only.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with persistent asthma.
* Not treated with the combination of a ICS (inhaled corticosteroid)and a LABA (long-acting beta-agonist).
* Female subjects must not be fertile or must use effective contraception.
* Subject must be able to comply with the use of the questionnaires in the local language.

Exclusion criteria:

* Known or suspected Chronic Obstructive Pulmonary Disease.
* Pregnant or lactating.
* Participating investigator, employee of an investigator, or family member of any of the aforementioned.
* Smoking history: Pack-years > 10 years.
* Have known clinical or laboratory evidence of a serious uncontrolled systemic disease.
* Known hypersensitivity to any substance contained in investigational product or as-needed medication.
* Treatment with oral corticosteroid within 2 months prior to the screening visit.
* Upper or lower respiratory tract infection (microbiologically verified) within 1 month prior to screening visit.
* Acute asthma exacerbation requiring hospitalisation or emergency room treatment within 3 months prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2005-07-26 (Actual); Primary Completion 2007-06-13 (Actual); Study Completion 2007-06-13 (Actual)

PRIMARY OUTCOMES:
number of subjects who achieved Total asthma Control: Period 2 | Up to Week 24
  Proportion of subjects who achieved Total Control in 7 out of the last 8 consecutive weeks in treatment period 2 with salmeterol/fluticasone propionate 50/250 g b.i.d. fixed dosing and compliance enhancement training compared with salmeterol/fluticasone propionate 50/250 g b.i.d. fixed dosing without compliance enhancement training.

SECONDARY OUTCOMES:
Number of subjects who achieved Total Control with salmeterol/fluticasone propionate 50/250 g b.i.d. fixed dosing: Period 2 | Up to Week 12
  Proportion of subjects who achieved Total Control with salmeterol/fluticasone propionate 50/250 g b.i.d. fixed dosing in treatment period 1 will be analyzed.
Time to first individual week with Total Control | Up to Week 24
  Time to first individual week with Total Control in treatment period 2 will be analyzed.
Morning peak expiratory flow (PEF) | Up to Week 24
  PEF is defined as a person's maximum speed of expiration and will be measured using a peak flow meter.
Forced expiratory volume in one second (FEV1) | Up to Week 24
  FEV1 is defined as Forced Expiratory Volume in the first second. The volume of air that can be forced out in one second after taking a deep breath, an important measure of pulmonary function.
Asthma symptom score | Up to Week 24
  Asthma symptom score will be analyzed to check the symptom severity
Number of subjects using rescue medication | Up to Week 24
  Rescue medication usage will be analyzed.
Number of nights with awakening due to asthma | Up to Week 24
  Number of nights with awakening due to asthma will be analyzed.
Asthma severity score | Up to Week 24
  Asthma severity score will be analyzed
Number of subjects with adverse events (AEs) | Up to Week 24
  Adverse events will be observed and counted.
AQLQ score | Up to Week 24
  Quality of life of subjects with asthma will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- Denmark (6):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Næstved
  - GSK Investigational Site, Odense C
- Switzerland (20):
  - GSK Investigational Site, Aarau
  - GSK Investigational Site, Allschwil
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Bever
  - GSK Investigational Site, Brittnau
  - GSK Investigational Site, Castione
  - GSK Investigational Site, Düdingen
  - GSK Investigational Site, Egg
  - GSK Investigational Site, Faltigberg-Wald
  - GSK Investigational Site, Horw
  - GSK Investigational Site, Klosters Platz
  - GSK Investigational Site, Malvaglia
  - GSK Investigational Site, Massagno
  - GSK Investigational Site, Pregassona
  - GSK Investigational Site, Steckborn
  - GSK Investigational Site, Thun
  - GSK Investigational Site, Wald
  - GSK Investigational Site, Wigoltingen
  - GSK Investigational Site, Worb

REFERENCES:
- [Derived] Ulrik CS, Claudius BK, Tamm M, Harving H, Siersted HC, Backer V, Hellquist B, Dahl R, Hogholm A, Johnk IK. Effect of asthma compliance enhancement training on asthma control in patients on combination therapy with salmeterol/fluticasone propionate: a randomised controlled trial. Clin Respir J. 2009 Jul;3(3):161-8. doi: 10.1111/j.1752-699X.2009.00129.x. PMID 20298399